CLINICAL TRIAL: NCT05978219
Title: Efficacy of Mirtazapine in Major Depressive Disorder With Insomnia: A 6-Week Pre and Post Intervention Study
Brief Title: Efficacy of Mirtazapine in Major Depressive Disorder With Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health, Dhaka (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Principal Investigator, Dr. Ahsan Aziz Sarkar, Co-investigator, National Institute of Mental Health, Dhaka
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/12
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder With Insomnia
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre-post intervention trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with MDD with insomnia (Experimental): Diagnosed MDD patients with insomnia problems will be approached and enrolled from NIMH, Dhaka.
  Trial medications will be self-administered and treatment regimen will be continued until serious adverse effect develops or for 42 days, whichever occurs sooner.
  Patients will receive mirtazapine at 15-30 mg/day (tablet form, once or twice daily, orally) from start. Depending on the response, doses might be increased at 2 weeks up to 45 mg/day for mirtazapine.
  The clinical trial for each patient will last for 42 days. Clinical data will be collected at the beginning - Day 0 and then on Day 14 and Day 42 of the trial by face-to-face interview. A clinical follow up will be provided to trial patients on Day 28 of the trial over telephone. Research psychiatrists will also conduct follow up, medication and side effect monitoring and overall management of the patients.
  Interventions: Drug: Mirtazapine Tablets

INTERVENTIONS:
Drug: Mirtazapine Tablets — Mirtazapine tablet form, orally, once or twice daily, 15-45 mg

SUMMARY:
This will be a single center, prospective, open label, quasi-experimental pre-post intervention trial in major depressive disorder (MDD) patients with insomnia.

The main objectives are i. to assess efficacy of mirtazapine in reducing depression and insomnia symptom severity in major depressive disorder (MDD) patients with insomnia.

ii. to evaluate side effects of mirtazapine.

Following enrollment and baseline assessment patients will be prescribed mirtazapine at 15-30 mg/day. Depending on the response, doses will be adjusted after two weeks and might be titrated up to 45 mg/day.

Each patient will be monitored for 42 days and assessment will be carried out on Day 0, Day 14, Day 28 and Day 42 of the trial.

DETAILED DESCRIPTION:
Background: Mirtazapine is an atypical antidepressant acts by increasing noradrenergic and serotonergic neurotransmission. It inhibits presynaptic adrenergic alpha-2 receptor along with inhibition of postsynaptic serotonergic 5-HT2 and 5-HT3 receptors and histamine (H1) receptor (Jilani et al., 2022). It was approved by FDA in 1996 for treating moderate and severe depression; but it also has sedative, antiemetic, anxiolytic, and appetite stimulant effects and for these prescribed in many other psychiatric disorders (Nutt, 2002). Because of its efficacy, safety and tolerability, it is one of the drugs recommended by NICE to consider as first-choice in treating depression (Middleton et al., 2005).

A depressive episode is characterized by a period of depressed mood or diminished interest in activities occurring most of the day, nearly every day during a period lasting at least two weeks accompanied by other symptoms such as difficulty concentrating, feelings of worthlessness or excessive or inappropriate guilt, hopelessness, recurrent thoughts of death or suicide, changes in appetite or sleep, psychomotor agitation or retardation, and reduced energy or fatigue. There have never been any prior manic, hypomanic, or mixed episodes, which would indicate the presence of a bipolar disorder (ICD-11, 2019).

Around 6.7% of adult population in Bangladesh suffers from depressive disorders (NIMH, 2019). However, no interventional study has yet been carried out to see efficacy of different antidepressants in this population. As one of the frequently observed features of depression is insomnia, mirtazapine could be a good choice in these cases. This study intends to assess the efficacy of mirtazapine in major depressive disorder when the patients also present with insomnia.

General objective To assess the efficacy of mirtazapine in reducing depression with insomnia symptoms in patients with major depressive disorder (MDD) with insomnia.

Specific objectives

1. To assess the efficacy of mirtazapine in reducing depressive symptoms in patients with MDD with insomnia.
2. To assess the efficacy of mirtazapine in reducing insomnia symptoms in patients with MDD with insomnia.
3. To compare the quality of life in patients with MDD before and after introducing mirtazapine.
4. To assess the side-effects experienced by trial patients.

Methods: This will be a single center, prospective, open label, quasi-experimental pre-post intervention trial in MDD patients with insomnia. The study will be conducted at National Institute of Mental Health (NIMH), Bangladesh over a period of 8 months. A total of 135 MDD patients with insomnia who fulfill the selection criteria will be conveniently selected for the study. Following enrollment and baseline assessment patients will be prescribed mirtazapine at 15-30 mg/day. Depending on the response, doses will be adjusted after two weeks and might be titrated up to 45 mg/day.

Each patient will be monitored for 42 days and assessment will be carried out on Day 0, Day 14, Day 28 and Day 42 of the trial. A semi-structured clinical information questionnaire, Hamilton Depression Rating Scale (HDRS), Insomnia Severity Index (ISI), Antidepressant Side-Effect Checklist (ASEC), World Health Organization Quality of Life (WHOQOL-BREF) will be used by research psychiatrists during assessment.

The whole study will be on accordance with Helsinki Declaration and prior to commencement, ethical approval will be taken from IRB and Bangladesh Medical Research Council (BMRC). The protocol will also be registered with the International Clinical Trials Registry Platform (ICTRP).

Potential significance: The findings will generate information on efficacy of mirtazapine in reducing depressive and insomnia symptom severity in MDD patients with insomnia and regarding side effects of mirtazapine in Bangladeshi adult population.

Funding: This study is conceptualized and sponsored by Bangladesh Association of Psychiatrists (BAP) with scientific support and research grant from Sun Pharmaceutical Bangladesh Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. Diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) for MDD.
3. A ≥20 total score on the 17-item Hamilton depression rating scale (HDRS).
4. A ≥15 total score on the 7-item Insomnia Severity Index (ISI).
5. Considered to require antidepressant treatment based on the judgment of the consulting psychiatrist.
6. For women - willing to abstain from conception or willing to use modern method of contraception (she or her partner) during trial period.

Exclusion Criteria:

1. History of use of mirtazapine in the last 3 months period.
2. Pregnant or breastfeeding mother.
3. At significant risk for suicide.
4. Diagnosed with a primary condition including dementia as well as bipolar, obsessive-compulsive, or eating disorders, schizophrenia, or alcohol or substance dependence except for tobacco dependence.
5. Experiencing any medical conditions judged to render the patient ineligible to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean Hamilton Depression Rating Scale score | At Day 0, Day 14 and Day 42
  Hamilton Depression Rating Scale is one of the most widely used clinician-administered depression assessment scale. The 17-item version score ranges between 0-53 with higher score indicates worse outcome.
Change from baseline in mean Insomnia Severity Index score | At Day 0, Day 14 and Day 42
  The Insomnia Severity Scale is a 7-item and 5-point Likert self-report questionnaire which is used to assess the nature, severity, and impact of insomnia. The total score can be between 0-35 and higher score indicates worse outcome.

SECONDARY OUTCOMES:
Frequency and severity of side effects experienced by trial patients as measured by Antidepressant Side-Effect Checklist | Day 14 and Day 42
  This is a self-reporting side-effect checklist developed by Royal College of the Psychiatrist for those taking antidepressants. There are 21 items each mentioning a particular side effect and for each item, the participants rated the severity of the specified symptom on a four-point scale (0 absent; 1 mild; 2 moderate; 3 severe) and specified whether a symptom (if present) was likely to be a side-effect of the antidepressant drug (yes or no).
Change from baseline in mean World Health Organization Quality of Life score | Day 0 and Day 42
  The WHOQOL-BREF is a 26-item questionnaire in a Likert scale format that assesses individuals' perceptions of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. The 26 items can be answered in a 1-5 Likert scale format; The scale is scored by adding up the score on each item to yield a total score for the instrument. It assesses quality of life in four domains namely physical, psychological, social and environmental. The converted scores for each domain range between 0-100 and a higher score indicates higher quality of life in that domain.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided